CLINICAL TRIAL: NCT00533377
Title: A Randomized, Placebo-Controlled Study To Evaluate The Efficacy, Safety And Tolerability Of CP-533,536 In Subjects With Closed Fracture Of The Tibial Shaft
Brief Title: ACTiF- Assessment of Closed Tibial Fractures
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A3241010
Record Dates: First submitted 2007-09-20; First posted 2007-09-21 (Estimated); Last update posted 2012-02-17 (Estimated); Status verified 2012-02

CONDITIONS: Tibial Fractures
MeSH Terms: conditions — Tibial Fractures | interventions — Standard of Care; CP533536

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- CP-533,536 Dose Level 2 (Experimental)
  Interventions: Drug: CP-533, 536
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Standard of Care (Other)
  Interventions: Procedure: Standard of Care
- CP-533,536 Dose Level 1 (Experimental)
  Interventions: Drug: CP-533,536
- CP-533,536 Dose Level 3 (Experimental)
  Interventions: Drug: CP-533,536
- CP-533.536 Dose Level 4 (Experimental)
  Interventions: Drug: CP-533,536

INTERVENTIONS:
Drug: CP-533, 536 — Active study drug
  Arms: CP-533,536 Dose Level 2
Drug: Placebo — Placebo vehicle
  Arms: Placebo
Procedure: Standard of Care — Standard surgical procedure
  Arms: Standard of Care
Drug: CP-533,536 — Active study drug
  Arms: CP-533,536 Dose Level 1
Drug: CP-533,536 — Active study drug
  Arms: CP-533,536 Dose Level 3
Drug: CP-533,536 — Active study drug
  Arms: CP-533.536 Dose Level 4

SUMMARY:
The purpose of this study is to find out the good and bad effects of an investigational drug called CP-533,536 in patients with closed fracture of the tibial shaft undergoing internal fixation using reamed inter-locked IM nailing procedure

ELIGIBILITY:
Inclusion Criteria:

* Males or females 17 years or older with confirmed closure of the tibial epiphyses, with a closed fracture of the tibial diaphysis undergoing treatment with reamed locked IM nailing procedure and the absence of an associated compartment syndrome or vascular injury;
* Closed tibial fractures Types A, B & C (See OTA fracture classification) can be included.

Exclusion Criteria:

* Previous fractures of the same tibia that may impact nailing procedure or impaired visibility of current fracture or a history of osteomyelitis;
* Subjects with any other clinically significant injuries, which may significantly impair weight bearing of the affected limb;
* Subjects with a fracture gap of >1cm after initial surgery and prior to drug administration;
* Any other planned invasive or non invasive interventions intended to promote bone healing of the tibial fracture under study are not allowed in the first 24 weeks after treatment.

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 276 (Actual)
Dates: Start 2008-01; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Time to fracture healing compared with placebo | 24 weeks

SECONDARY OUTCOMES:
Proportion of subjects who require a secondary intervention to promote fracture healing | 48 weeks
Impact on the subject's ability to return to normal function, general health status, work productivity, and degree of pain at fracture site compared with placebo and Standard of Care groups | 24 weeks
Time to fracture healing compared with Standard of Care | 24 weeks
Proportion of patients healed compared with placebo | 16 weeks
Time to regular callus formation compared with placebo | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (45):
- United States (10):
  - Pfizer Investigational Site, Wichita, Kansas
  - Pfizer Investigational Site, Worcester, Massachusetts
  - Pfizer Investigational Site, Minneapolis, Minnesota
  - Pfizer Investigational Site, Columbia, Missouri
  - Pfizer Investigational Site, Durham, North Carolina
  - Pfizer Investigational Site, Chattanooga, Tennessee
  - Pfizer Investigational Site, Dallas, Texas
  - Pfizer Investigational Site, Houston, Texas
  - Pfizer Investigational Site, Salt Lake City, Utah
  - Pfizer Investigational Site, Morgantown, West Virginia
- Australia (2):
  - Pfizer Investigational Site, Herston, Queensland
  - Pfizer Investigational Site, Adelaide, South Australia
- Pfizer Investigational Site, Sarajevo, Bosnia and Herzegovina
- Canada (6):
  - Pfizer Investigational Site, Red Deer, Alberta
  - Pfizer Investigational Site, Hamilton, Ontario
  - Pfizer Investigational Site, London, Ontario
  - Pfizer Investigational Site, Ottawa, Ontario
  - Pfizer Investigational Site, Sarnia, Ontario
  - Pfizer Investigational Site, Toronto, Ontario
- Croatia (2):
  - Pfizer Investigational Site, Varaždin
  - Pfizer Investigational Site, Zagreb
- India (6):
  - Pfizer Investigational Site, Secunderabad, Andhra Pradesh
  - Pfizer Investigational Site, Bangalore, Karnataka
  - Pfizer Investigational Site, Mangalore, Karnataka
  - Pfizer Investigational Site, Mumbai, Maharashtra
  - Pfizer Investigational Site, Ludhiana, Punjab
  - Pfizer Investigational Site, Lucknow, Uttar Pradesh
- Japan (9):
  - Pfizer Investigational Site, Nagoya, Aichi-ken
  - Pfizer Investigational Site, Kitakyushu-shi, Fukuoka
  - Pfizer Investigational Site, Mizumaki-cho Onga-gun, Fukuoka
  - Pfizer Investigational Site, Okawa-shi, Fukuoka
  - Pfizer Investigational Site, Fujisawa-shi, Kanagawa
  - Pfizer Investigational Site, Kouchi, Kouchi-ken
  - Pfizer Investigational Site, Sasebo-Shi, Nagasaki
  - Pfizer Investigational Site, Toda-shi, Saitama
  - Pfizer Investigational Site, Shinagawa-ku, Tokyo
- Pfizer Investigational Site, Saint Petersburg, Russia
- South Africa (4):
  - Pfizer Investigational Site, Parktown, Gauteng
  - Pfizer Investigational Site, Glenwood, KwaZulu-Natal
  - Pfizer Investigational Site, Soweto
  - Pfizer Investigational Site, Tygerberg
- Pfizer Investigational Site, Seville, Sevilla, Spain
- Turkey (Türkiye) (3):
  - Pfizer Investigational Site, Ankara
  - Pfizer Investigational Site, Istanbul
  - Pfizer Investigational Site, Izmir

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3241010&StudyName=ACTiF-%20Assessment%20of%20Closed%20Tibial%20Fractures